CLINICAL TRIAL: NCT04500158
Title: The Effect of Local Anesthesia When Used in Dental Restorative Cases Under General Anesthesia on Control of Intraoperative Physiologic Parameters and Post Operative Comfort
Brief Title: The Effect of Local Anesthesia on Control of Intraoperative Physiologic Parameters and Post Operative Comfort
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: HM20018316
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Pain, Procedural
MeSH Terms: conditions — Pain, Procedural | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Local anesthesia (Experimental): Participants will receive local anesthesia in addition to the standard care general anesthesia
  Interventions: Drug: Lidocaine
- Standard care (No Intervention): Participants will receive standard care general anesthesia

INTERVENTIONS:
Drug: Lidocaine — 2% Lidocaine with 1:100,000 epi
  Arms: Local anesthesia

SUMMARY:
The purpose of this study is to compare patient responses during and after surgery when local anesthetic is used for dental treatment under general anesthesia (GA) and when it is not used.

DETAILED DESCRIPTION:
Local anesthesia is a widely used tool to ensure patient safety and comfort in the dental office. This is usually accomplished by administering a shot of numbing medicine (local anesthesia) in different parts of the mouth. Local anesthesia is an important tool used for care in the dental office however despite its standardized use in dental clinics use of local anesthetic is not standardized for use in dental cases under GA. In the literature there is some evidence suggesting that it has some marginal benefit for pain control short term post operatively and control of vital signs during surgery. Some evidence also suggests that due to its use there can be increase in post-operative lip chewing and cheek biting due to the numb sensation. Additionally, it has been seen that due to the numb sensation that children can be more irritable during when waking up after surgery.

The study section will have 60 participants of which one half will receive local anesthesia for restorative dental care under GA and the other half will receive conventional no anesthesia for restorative dental treatment under GA, based on random assignment (like the flip of a coin). There is an equal chance of being assigned to either group prior to the consented treatment. Before the surgery, a nurse will access the child's overall pain and comfort. The study team (faculty, anesthesiologist, and resident) will record the blood pressure, heart rate, and breathing duration throughout the procedure. After the child has completed the surgery a nurse will again access the child's overall pain and comfort. Lastly, parents will be contacted that evening of surgery by a member of the study team to check up on the child and will be asked some questions to access the child's comfort at home.

ELIGIBILITY:
Inclusion Criteria:

• Pediatric patients undergoing GA for dental restorative work at Virginia Commonwealth University Children's Hospital of Richmond Pavilion and Brook Road Centers

Exclusion Criteria:

* Children with any sensory or behavioral issues
* Patients requiring extractions or surgical procedures

Max Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2020-11-03 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Bortell, DDS, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Local Anesthesia | Standard Care
Started | 32 | 27
Completed | 15 | 16
Not Completed | 17 | 11
Not completed — Physician Decision | 17 | 11

BASELINE CHARACTERISTICS:
Population: Number of subjects that completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Local Anesthesia | Standard Care | Total
Number analyzed (Participants) | 15 | 16 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 16 | 31
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 9 | 10 | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 1 | 6
  Not Hispanic or Latino | 10 | 15 | 25
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 11 | 16
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 3 | 10

OUTCOME MEASURES:

1. Primary Outcome: Post Operative Pain
Description: The Parent's Postoperative Pain Measure ( abbreviated: PPPM) Scale consists of 15 questions with scores ranging from 0 to 15, with one point assigned to each question answered with a "Yes" and therefore higher scores indicating worse postoperative pain. A score of 6 or greater is considered clinically significant pain which was tallied for the primary outcome measure (i..e number of participants experiencing clinically significant postoperative pain).
Time Frame: in the evening of the day of surgery, up to 10 hours
Population: Number of parents that completed the parents post operative pain measure
Measure: Count of Participants; unit: Participants
Arm/Group | Local Anesthesia | Standard Care
Number analyzed (Participants) | 15 | 16
Participants | 13 | 10

2. Secondary Outcome: Number of Teeth Treated
Description: Will report the mean and standard deviation of number of teeth treated
Time Frame: start of procedure to end of procedure, the intraoperative time frme
Population: Number of subjects that completed the study.
Measure: Mean (Standard Deviation); unit: teeth treated
Arm/Group | Local Anesthesia | Standard Care
Number analyzed (Participants) | 15 | 16
teeth treated | 8.6 (3.4) | 7.4 (3.4)

3. Secondary Outcome: Procedure Time
Description: Will report the mean and standard deviation of the procedure time
Time Frame: start of procedure to end of procedure, minutes
Population: Number of subjects that completed the study.
Measure: Mean (Standard Deviation); unit: procedure time in minutes
Arm/Group | Local Anesthesia | Standard Care
Number analyzed (Participants) | 15 | 16
procedure time in minutes | 85.4 (32.8) | 70.6 (29)

4. Secondary Outcome: PACU Time
Description: Will report the mean and standard deviation of time after the procedure to through time in the post-anesthesia care unit
Time Frame: time from after procedure to through time in the post-anesthesia care unit in minutes
Population: Number of subjects that completed the study
Measure: Mean (Standard Deviation); unit: Time in minutes
Arm/Group | Local Anesthesia | Standard Care
Number analyzed (Participants) | 15 | 16
Time in minutes | 39.8 (11.6) | 39.9 (9.3)

ADVERSE EVENTS:
Time Frame: Subjects were followed for the day of the procedure
Arm/Group | Local Anesthesia | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT04500158/Prot_SAP_001.pdf
  • Informed Consent Form (2022-12-01): https://cdn.clinicaltrials.gov/large-docs/58/NCT04500158/ICF_002.pdf